CLINICAL TRIAL: NCT07282574
Title: A Multi-center, Double-blind, Placebo-controlled, Phase II Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of RO7268489, a Monoacylglycerol Lipase Inhibitor, as Add-on Therapy to Ocrelizumab, in Participants With Progressive Forms of Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of RO7268489 as Add-on Therapy to Ocrelizumab, in Participants With Progressive Forms of Multiple Sclerosis (MS)
Acronym: Mintaka
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP46016; 2025-521636-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RO7268489 Dose 1 + Ocrelizumab (Experimental): Participants will receive RO7268489 along with ocrelizumab as per the pre-defined regimen.
  Interventions: Drug: RO7268489; Drug: Ocrelizumab
- RO7268489 Dose 2 + Ocrelizumab (Experimental): Participants will receive RO7268489 along with ocrelizumab as per the pre-defined regimen.
  Interventions: Drug: RO7268489; Drug: Ocrelizumab
- RO7268489 Dose 3 + Ocrelizumab (Experimental): Participants will receive RO7268489 along with ocrelizumab as per the pre-defined regimen.
  Interventions: Drug: RO7268489; Drug: Ocrelizumab
- Placebo + Ocrelizumab (Placebo Comparator): Participants will receive RO7268489 matching placebo along with ocrelizumab as per the pre-defined regimen.
  Interventions: Drug: Ocrelizumab; Drug: Placebo

INTERVENTIONS:
Drug: RO7268489 — RO7268489 will be administered per schedule as specified in the arms.
  Arms: RO7268489 Dose 1 + Ocrelizumab; RO7268489 Dose 2 + Ocrelizumab; RO7268489 Dose 3 + Ocrelizumab
Drug: Ocrelizumab — Ocrelizumab will be administered per schedule as specified in the arms.
  Other Names: RO4964913, Ocrevus
Drug: Placebo — Placebo will be administered per schedule as specified in the arms.
  Arms: Placebo + Ocrelizumab

SUMMARY:
The main purpose of this study is to assess the efficacy of RO7268489 in adults with progressive multiple sclerosis (PMS) receiving ocrelizumab. After the end of the double-blind period, an open-label (OL) extension may allow eligible participants to receive open-label RO7268489.

ELIGIBILITY:
Inclusion Criteria:

* PMS, in accordance with the revised 2017 McDonald criteria
* Expanded disability status scale (EDSS) at screening between 3.0 and 6.0 inclusive

Exclusion Criteria:

* MS relapse during the 6 months preceding the randomization date
* Lack of peripheral venous access
* History of alcohol or other drug abuse, in the opinion of the investigator, within 5 years prior to screening
* Inability to complete an magnetic resonance imaging (MRI)
* Contraindications to ocrelizumab mandatory pre-medications
* Treatment with intravenous immunoglobulin (IV Ig) or plasmapheresis within 12 weeks prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Time From Randomization to the First Occurrence of Composite Confirmed Disability Progression (cCPD) Confirmed for at Least 12 Weeks (cCDP12) | Up to approximately 110 weeks
  Time from randomization to the first occurrence of cCDP12 according to at least one of the following 3 criteria:
  1. 12-week confirmed disability progression (CDP12)
  2. 12-week confirmed increase in Timed 25-Foot Walk Test (T25FWT) or
  3. 12-week confirmed increase in 9-Hole Peg Test (9-HPT) The EDSS is a disability scale is based on a standard neurological examination that ranges in 0.5-point steps from 0 (normal) - 10 (death). T25FWT=time taken to walk 25 feet, typically measured in seconds. The longer it takes to walk, the higher score, which indicates deterioration. Lower times indicate better performance and greater mobility. In 9-HPT, participants are instructed to place pegs one by one into each of nine holes arranged in a board stabilized with a plastic nonslip sheet on a solid table, and then to remove these pegs from the holes. The shorter time it takes to complete the task indicates a better outcome.

SECONDARY OUTCOMES:
Time From Randomization to the First Occurrence of 24-Week Confirmed ≥4-Point Decrease (Worsening) in Symbol Digit Modalities Test (SDMT) | Up to approximately 110 weeks
  The SDMT is a performance measure of processing speed that is widely used to assess cognitive function in response to treatment. It's brief, easy to administer, and involves a simple substitution task that healthy children and adults can easily perform. Using a reference key, the participant has 90 seconds to pair specific numbers with given geometric figures. The total SDMT score is the total number of correct responses and ranges from 0 to 110, with a higher score indicating a higher level of processing speed. A four-point change from baseline is typically considered clinically meaningful.
Change From Baseline in Total Brain Volume | Up to approximately 110 weeks
Time to Onset of 24-Week cCDP (cCDP24) | Up to approximately 110 weeks
Time to Onset of 12-Week Confirmed Disability Progression CDP (CDP12) | Up to approximately 110 weeks
Time to Onset of 24-Week CDP (CDP24) | Up to approximately 110 weeks
Time to ≥ 20% Increase in 12-week Confirmed Timed 25-Foot Walk Test (T25FWT) | Up to approximately 110 weeks
  The time taken to walk 25 feet, typically measured in seconds. The longer it takes to walk, higher the score, which indicates deterioration and greater impairment. Lower times indicate better performance and greater mobility. Lower the mean change in the score over time, the better performance.
Time to ≥ 20% Increase in 24-week Confirmed T25FWT | Up to approximately 110 weeks
  The time taken to walk 25 feet, typically measured in seconds. The longer it takes to walk, higher the score, which indicates deterioration and greater impairment. Lower times indicate better performance and greater mobility. Lower the mean change in the score over time, the better performance.
Time to ≥ 20% Increase in 12-week Confirmed 9-Hole Peg Test (9-HPT) | Up to approximately 110 weeks
  Participants are instructed to place pegs one by one into each of nine holes arranged in a board stabilized with a plastic nonslip sheet on a solid table, and then to remove these pegs from the holes. Both the dominant and non-dominant hands are tested twice (two consecutive trials for each hand). The participants are required to complete two successful trials for each hand. The amount of time (in seconds) required to place and remove all nine pegs is recorded for each trial. More time = higher raw scores, which indicates deterioration. The lower mean change in the score over time, the better the performance.
Time to ≥ 20% Increase in 24-week Confirmed 9-HPT | Up to approximately 110 weeks
  Participants are instructed to place pegs one by one into each of nine holes arranged in a board stabilized with a plastic nonslip sheet on a solid table, and then to remove these pegs from the holes. Both the dominant and non-dominant hands are tested twice (two consecutive trials for each hand). The participants are required to complete two successful trials for each hand. The amount of time (in seconds) required to place and remove all nine pegs is recorded for each trial. More time = higher raw scores, which indicates deterioration. The lower mean change in the score over time, the better the performance.
Plasma 2-arachidonoylglycerol (2-AG) Levels | Up to approximately 110 weeks
Change From Baseline in Plasma 2-AG Levels | Up to approximately 110 weeks
Number of Participants With Adverse events (AEs) | Up to 5 years
Number of Participants With Treatment Discontinuations due to AEs | Up to 5 years
Proportion of Participants With Suicidal Ideation or Behavior, as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 5 years
  C-SSRS is an assessment tool used to assess lifetime suicidality of participant (at baseline) as well as any new instances of suicidality (C-SSRS since last visit). Structured interview prompts recollection of suicidal ideation, including intensity of ideation, behavior, and attempts with actual/potential lethality. Categories have binary responses (yes/no) and include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior is indicated by a "yes" answer to any of the listed categories. Score of 0 is assigned if no suicide risk is present. Score of 1 or higher indicate suicidal ideation or behavior.
Plasma Concentrations of RO7268489 and Its Metabolite(s) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University of Medicine, Ankara
  - Gazi University Medical Faculty, Ankara

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing